CLINICAL TRIAL: NCT01358136
Title: ThyrOp: Individual Subclinical Hypothyroidism After Hemithyroidectomy for Benign Nontoxic Goiter - Focus on Weight Gain and Mitochondrial Dysfunction
Brief Title: ThyrOp: A Study of Individual Subclinical Hypothyroidism After Hemithyroidectomy for Benign Nontoxic Goiter
Acronym: ThyrOp
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Naestved Hospital (Other)
Collaborators: Denmark:Department of Otorhinolaryngology Slagelse Hospital, Hospital South (Unknown); Region Zealand (Other)
Responsible Party: Principal Investigator, Tina Toft Kristensen, Ph.D Student, MD, Naestved Hospital
Other Study IDs: SJ-10
Record Dates: First submitted 2011-05-18; First posted 2011-05-23 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Goiter; Hypothyroidism; Weight Gain
Keywords: Thyroidectomy; Mitochondria
MeSH Terms: conditions — Goiter; Hypothyroidism; Weight Gain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hemithyroidectomy: Patients with benign nontoxic goiter who have an indication for hemithyroidectomy

SUMMARY:
The hypothesis of the study is that among patients that do not develop overt hypothyroidism after hemithyroidectomy, weight gain is a clinical manifestation of a postoperatively lowered set point of thyroid function - even if the thyroid function is lowered within the laboratory reference range. The investigators refer to this hypothesized condition as individual subclinical hypothyroidism.

Thyroid hormones are major regulators of mitochondrial function and subclinical hypothyroidism affects mitochondrial activity. The aim of the study is to examine if a lowered set point of thyroid function after hemithyroidectomy can be measured in the mitochondrial function, the body weight and the basal oxygen consumption.

DETAILED DESCRIPTION:
The operation of hemithyroidectomy (total thyroid lobectomy and isthmusectomy with preservation of the contralateral lobe) is indicated for patients with a unilateral thyroid mass that is causing compressive symptoms, cosmetic concern or to exclude thyroid carcinoma.

The incidence and risk factors for development of hypothyroidism after hemithyroidectomy remain unclear. The reported rates of postoperative hypothyroidism vary from 5.0% to 41.9 % because of variable follow-up and definition of hypothyroidism (Wormald et al). There are no nationally nor universally accepted guidelines for the monitoring of thyroid function after hemithyroidectomy.

Subclinical hypothyroidism is associated with an increased risk of coronary heart events and coronary heart mortality (Rodondi et al) and a high level of thyrotropin (within the laboratory reference range) has been related to an increased risk of fatal coronary heart disease (Asvold et al) Variation in thyroid function is seen between individuals also within the normal range. The individual variation in serum levels of thyroid hormones and thyrotropin between measurements in the same individual is relatively small compared with variations between individuals (Andersen et al). This implicates that around half of the laboratory reference range for thyrotropin is abnormal for a given individual. The fact that a thyrotropin value of an individual can be within the reference range but still represent an abnormal thyroid function in that given person has consequences for the monitoring of thyroid function after hemithyroidectomy. It implies that the postoperative thyroid function should be monitored by having the preoperative thyroid function in mind and that postoperative hypothyroidism should be understood in a broader term. After hemithyroidectomy a change in the individual unique set point that results in a lowered thyroid function can represent a condition that the investigators refer to as individual subclinical hypothyroidism.

Weight gain following hemithyroidectomy for benign nodular goiter among patients that do not develop overt hypothyroidism is a frequent clinical observation. Body weight is influenced by many factors, there among thyroid function. Even small differences in thyroid function with s-thyrotropin variations within the normal laboratory range for patients on T4 substitution therapy are associated with differences in resting energy expenditure. A prolonged decrease in REE could lead to increased body weight (al-Adsani et al).

Overweight and obesity are major threats to public health. The importance of lifestyle for weight gain is not to be doubted but other factors such as slight differences in thyroid function might be of importance in the risk of gaining weight as well (Knudsen et al).

The mitochondria provide cellular energy by converting oxygen and nutrients into ATP by aerobe respiration and mitochondrial energy production is regulated by thyroid hormones (Weitzel et al). Subclinical hypothyroidism has previously been shown to affect mitochondrial function in mononuclear blood cells (Kvetny et al).

The investigators hypothesize that after hemithyroidectomy some patients develop lowered thyroid function which results in a postoperative higher value of serum thyrotropin as a consequence of less negative feed-back on the pituitary gland. Weather the postoperative lowered thyroid function results in overt hypothyroidism (serum thyrotropin above the upper reference limit, lowered serum levels of free T3 and T4), subclinical (serum thyrotropin above the upper reference limit, free T3 and T4 within the reference range) or individual subclinical hypothyroidism (serum thyrotropin rises within the reference range, free T3 and T4 within the reference range) depends on the preoperative set point of thyroid function of the given patient but either condition represents a condition that is abnormal. The investigators hypothesize that a postoperative lowered thyroid function will affect mitochondrial function and result in weight gain.

ELIGIBILITY:
Inclusion Criteria:

* Is going to undergo hemithyroidectomy for nontoxic goiter at the department of otorhinolaryngology at Slagelse Hospital, Denmark.
* BMI 20-40
* No past thyroid diseases
* No medication with influence on the pituitary-thyroid axis
* No hormone replacement therapy
* No childbirth or pregnancy within the last year
* Not currently breastfeeding

Exclusion Criteria:

* Malignant goiter, diagnosed by histological examination of the resected tissue
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is patients who meet the inclusion criteria and who are going to undergo hemithyroidectomy at Slagelse Hospital in Region Zealand, Denmark. The study subjects are are invited to participate by letter after the operation date is been scheduled.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-08 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Change in mitochondrial function from baseline value (before hemithyroidectomy) | 12 months after hemithyroidectomy
  Mitochondrial function is examined by 1) measurement of mitochondrial mass and mitochondrial membrane potential by flow cytometry and by 2) examination of expression of mitochondrial-related genes measured by real time PCR.

SECONDARY OUTCOMES:
Change in body weight and body composition from baseline value (before hemithyroidectomy) | 12 months after hemithyroidectomy
  Body weight and body composition is measured by weight in kilograms and by bioelectrical impedance analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Slagelse Hospital, Hospital South, Slagelse, Region Sjælland, Denmark

REFERENCES:
- [Background] Kvetny J, Wilms L, Pedersen PL, Larsen J. Subclinical hypothyroidism affects mitochondrial function. Horm Metab Res. 2010 May;42(5):324-7. doi: 10.1055/s-0030-1248261. Epub 2010 Feb 22. PMID 20178065
- [Background] Wormald R, Sheahan P, Rowley S, Rizkalla H, Toner M, Timon C. Hemithyroidectomy for benign thyroid disease: who needs follow-up for hypothyroidism? Clin Otolaryngol. 2008 Dec;33(6):587-91. doi: 10.1111/j.1749-4486.2008.01794.x. PMID 19126134
- [Background] Andersen S, Pedersen KM, Bruun NH, Laurberg P. Narrow individual variations in serum T(4) and T(3) in normal subjects: a clue to the understanding of subclinical thyroid disease. J Clin Endocrinol Metab. 2002 Mar;87(3):1068-72. doi: 10.1210/jcem.87.3.8165. PMID 11889165
- [Background] al-Adsani H, Hoffer LJ, Silva JE. Resting energy expenditure is sensitive to small dose changes in patients on chronic thyroid hormone replacement. J Clin Endocrinol Metab. 1997 Apr;82(4):1118-25. doi: 10.1210/jcem.82.4.3873. PMID 9100583
- [Background] Knudsen N, Laurberg P, Rasmussen LB, Bulow I, Perrild H, Ovesen L, Jorgensen T. Small differences in thyroid function may be important for body mass index and the occurrence of obesity in the population. J Clin Endocrinol Metab. 2005 Jul;90(7):4019-24. doi: 10.1210/jc.2004-2225. Epub 2005 May 3. PMID 15870128
- [Background] Weitzel JM, Iwen KA, Seitz HJ. Regulation of mitochondrial biogenesis by thyroid hormone. Exp Physiol. 2003 Jan;88(1):121-8. doi: 10.1113/eph8802506. PMID 12552316
- [Background] Rodondi N, den Elzen WP, Bauer DC, Cappola AR, Razvi S, Walsh JP, Asvold BO, Iervasi G, Imaizumi M, Collet TH, Bremner A, Maisonneuve P, Sgarbi JA, Khaw KT, Vanderpump MP, Newman AB, Cornuz J, Franklyn JA, Westendorp RG, Vittinghoff E, Gussekloo J; Thyroid Studies Collaboration. Subclinical hypothyroidism and the risk of coronary heart disease and mortality. JAMA. 2010 Sep 22;304(12):1365-74. doi: 10.1001/jama.2010.1361. PMID 20858880
- [Background] Asvold BO, Bjoro T, Nilsen TI, Gunnell D, Vatten LJ. Thyrotropin levels and risk of fatal coronary heart disease: the HUNT study. Arch Intern Med. 2008 Apr 28;168(8):855-60. doi: 10.1001/archinte.168.8.855. PMID 18443261